CLINICAL TRIAL: NCT04481386
Title: A Phase I, Safety and Tolerability Study of Vitargus® in Vitrectomy Surgery
Brief Title: A Phase I Study of Vitargus® in Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioFirst Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFC-1401
Record Dates: First submitted 2020-07-15; First posted 2020-07-22 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Vitreo-retinal Surgery

STUDY DESIGN:
Intervention Model Description: A single intravitreal (IVT) dose of BFC-1401 in participants as a vitreous substitute during vitrectomy surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active arm (Experimental): Participants with a diagnosis of retinal detachment or vitreous haemorrhage, who are scheduled for vitrectomy surgery with a vitreous substitute
  Interventions: Device: Vitargus, BFC-1401

INTERVENTIONS:
Device: Vitargus, BFC-1401 — A single intravitreal (IVT) dose of BFC-1401 in participants as a vitreous substitute during vitrectomy surgery.

SUMMARY:
A Phase I, safety and tolerability study of Vitargus® in vitrectomy surgery

DETAILED DESCRIPTION:
Study Objectives:

Primary Objective

• To evaluate the safety/tolerability of a single intravitreal (IVT) dose of BFC-1401 in participants as a vitreous substitute during vitrectomy surgery.

Secondary Objective

* To assess retinal attachment and hydrogel degradation at Day 120.
* To assess best corrected visual acuity (BCVA) after vitrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, aged 18 years or older at screening.
2. a) Diagnosis of Diagnosis of Diagnosis of Diagnosis of complex or rhegmatogenous retinal detachment, or chronic retinal detachment with failure of gas or silicone oil treatment, OR b) Diagnosis of any vitreous haemorrhage that requires vitrectomy surgery
3. BCVA of 20/40 to 20/2000.
4. Scheduled vitrectomy with vitreous substitute.
5. Must be able and willing to provide written informed consent, attend all scheduled visits and comply with all study procedures.

Exclusion Criteria:

A participant meeting any of the following criteria was to be excluded from the study:

1. Any active intraocular or periocular infection or inflammation.
2. Only one functional eye.
3. Ocular disorders in the study eye that may confound the interpretation of the study results; macular oedema not requiring vitrectomy surgery, choroidal neovascularisation.
4. High refractive error demonstrating >6 diopters of myopia.
5. Any ophthalmic condition that reduces the clarity of the optical media that interferes with ophthalmic examination and adequate imaging (advanced cataract or corneal opacities).
6. Uncontrolled glaucoma defined as intraocular pressure > 30 mmHg on maximal therapy.
7. Aphakia or absence of the posterior capsule.
8. Known hypersensitivity to hyaluronic acid or ADH.
9. Uncontrolled blood pressure defined as systolic value ≥ 160 mmHg or diastolic value ≥100 mmHg at screening.
10. Uncontrolled diabetes defined as glycated haemoglobin (HbA1c) > 12%.
11. Stroke or myocardial infarction within 90 days of baseline.
12. Severe generalised disease resulting in a life expectancy shorter than 1 year.
13. Currently pregnant or breastfeeding.
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment. Effective contraception methods included:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) was not acceptable.
    * Female sterilisation (surgical bilateral oopthorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, this was acceptable only when the reproductive status of the woman was confirmed by follow-up hormone level assessment.
    * Male sterilisation (at least 6 months prior to screening). For female participants on the study, the vasectomised male partner was to be the sole partner for that participant.
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate<1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Placement of an intrauterine device or intrauterine system.
    * In the case of use of oral contraception, women were to be stable on the same pill for a minimum of 3 months before taking study treatment.
    * The use of an effective contraception method was to continue for 4 months post-vitrectomy and injection of the investigational product, in line with the follow-up period of the study.
    * Because the experimental investigational product in this study may affect an unborn baby, males participating in this study were not to father a baby while on the study, and for 4 months following the injection of study medication.
    * Women were considered post-menopausal and not of child-bearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation, at least six weeks prior to the study. In the case of oophorectomy alone, only when the reproductive status of the woman was confirmed by follow-up hormone level assessment was she considered to be not of child-bearing potential.
15. Participation in any study involving an investigational drug or device within the past 30 days or ongoing participation in a study with an investigational drug or device.
16. Any clinical evidence that the Investigator felt would place the participant at increased risk with the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability: Incidence of Treatment-Emergent Adverse Events | 120 days
  Incidence of Treatment-Emergent Adverse Events. Adverse events (AEs) were coded using the Medical Dictionary for Regulatory Activities (MedDRA), and data summarised by System Organ Class and preferred term.

SECONDARY OUTCOMES:
Efficacy for best corrected visual acuity (BCVA); retinal attachment and hydrogel degradation | 120 days
  To assess best corrected visual acuity (BCVA) by LogMAR change from baseline over time after vitrectomy surgery.
  To assess retinal attachment and hydrogel degradation by slit lamp biomicroscopy exam findings, dilated ophthalmoscopy exam findings, colour fundus photography, and OCT findings over time after vitrectomy surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, MD, Ph.D, Principal Investigator — Sydney Retina Clinic | Medical Director
Locations (1):
- Sydney Retina Clinic and Day Surgery, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.globenewswire.com/news-release/2019/10/15/1930092/0/en/American-BriVision-Highlights-Results-from-Vitargus-First-in-Human-Clinical-Trial.html